CLINICAL TRIAL: NCT04653896
Title: Design Improvements and Evaluation of a Knee Stress-Relief Powered Exoskeleton for Veterans With Knee Osteoarthritis
Brief Title: A Powered Exoskeleton for Veterans With Knee OA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: VA Pittsburgh Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A3228-R; RX-003228-01A2 (Other: VA R&D Merit Review)
Record Dates: First submitted 2020-11-12; First posted 2020-12-04 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Knee Osteoarthritis
Keywords: knee; arthritis; walking
MeSH Terms: conditions — Osteoarthritis, Knee; Arthritis

STUDY DESIGN:
Intervention Model Description: We will conduct a functional mobility comparison between Keeogo and knee braces among participants with knee OA. A within-subject design is selected. We plan to have 2 or 3 1-hour sessions per week (up to 12 sessions) for tuning the Keeogo and letting the participants be familiar with the device. After that, participants will be evaluated through a series of mobility tests using their prescribed knee braces and Keeogo configured with tuned parameters, respectively. If participants can complete the mobility tests without their knee braces we will also collect these data. The functional mobility tests will include the 6 Minute Walk Test, Timed Up and Go, 13-step Stair Test, Pick up Penny from Floor Test, and Short Physical Performance Battery. The investigators expect to use two separate sessions to finish the evaluations. The order of using the Keeogo and their knee braces will be randomized. There will be a 10-min break between each test. Participants could request a longer break time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Knee OA group (Experimental): Individuals who are over 18 years and have medical diagnosis of Grade 3 or 4 knee OA
  Interventions: Device: Keeogo

INTERVENTIONS:
Device: Keeogo — The Keeogo is the only commercially available (in Canada) robotic exoskeleton for a non-paralyzed population who can stand and initiate a stepping action, but have impaired mobility for functional tasks. Keeogo provides active assistance during stance and swing phases and assists users to perform functional mobility tasks including walking, stair climbing, sit-to-stand, bending, squatting, and kneeling.

SUMMARY:
The purpose of this study is to evaluate in-laboratory mobility outcomes, pain perception, and user satisfaction with the Keeogo , a robotic exoskeleton for providing assistance on knees during stand and swing for a population with impaired mobility, as compare with standard knee braces. The investigators hypothesize that participants could have improved performance outcomes on walk test, timed up and go test, stair test, pick up penny from floor test, and the Short Physical Performance Battery (SPPB) when using the Keeogo as compared with their prescribed knee braces.

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) is a growing problem due to increased longevity and obesity with estimates of 14 million people living with this impairment. Knee OA results in decreased activity and lifestyle changes, further exacerbating an individual's health. Exoskeleton technology (Keeogo , B-temia, Inc.) may be a viable alternative to standard knee OA treatment by providing powered support to reduce pain during mobility. To the investigators' knowledge, the Keeogo is the only commercially available (in Canada) robotic exoskeleton for a non-paralyzed population who can stand and initiate a stepping action, but have impaired mobility for functional tasks. Keeogo provides active assistance during stance and swing phases and assists users to perform functional mobility tasks including walking, stair climbing, sit-to-stand, bending, squatting, and kneeling. Preliminary studies with the Keeogo in six persons with knee OA showed efficacy for pain reduction during different mobility tasks. Keeogo may have the potential to address functional mobility problems and pain in Veterans with knee OA but is not yet approved by the FDA. An in-laboratory evaluation of performance outcomes using the Keeogo compared with standard knee braces are lacking. Absence of published prescription and general guidelines for use in Veterans with knee OA were also identified as limitations.

The purpose of this study is to evaluate in-laboratory mobility outcomes, pain perception, and user satisfaction with the Keeogo as compare with standard knee braces. The investigators hypothesize that participants could have improved performance outcomes on mobility tests, including a 6-minute walk test, timed up and go test, 13-step stair test, pick up penny from floor test, and the Short Physical Performance Battery (SPPB) when using the Keeogo as compared with their prescribed knee braces and reduced pain with the Keeogo by the numeric pain rating scale (NPRS) as compared with their prescribed knee braces for the mobility tests.

A knee OA-specific tuning protocol will be developed and used in the in-laboratory evaluations in 26 Veterans with knee OA at the James J. Peters VA Medical Center, Bronx, NY. This in-laboratory study is expected to demonstrate improved walking velocities, stair ascent/descent times, improved sit-to-stand, stand-to-sit, and object retrieval from the floor with reduced pain while participants use the Keeogo.

ELIGIBILITY:
Inclusion Criteria:

* medical diagnosis of Grade 3 or 4 knee OA
* have a prescribed knee brace for at least three months
* self-reported knee pain when standing, walking, climbing stairs, squatting, or other mobility activities
* self-reported limitations to mobility and walking activities due to knee pain, stiffness, loss of range of motion

Exclusion Criteria:

* neurological paralysis causing an inability to stand, weight bear or take stepping movements
* fixed contractures resulting in limited range of motion in the hip, knees, or ankles that prevent sitting, standing, walking, and/or squatting activities
* able to walk at a normal walking speed (>1.2 m/s) based on a 6-minute walk test (6MWT)
* anthropometric incompatibility with the device
* any medical complication or co-morbidity as judged by the study physician to be contraindicated for wearing the device or walking (e.g., cardiovascular disorders, pressure ulcers, open wounds, lower limb vascular disorders, or other medical conditions)
* a score of <8/10 on the MacArthur Competence Assessment Tool for Treatment (MacCAT-T) (as a proxy for cognitive competency screening); and 7) pregnancy or planning on becoming pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Changes of 6-Minute Walk Test results among different conditions | Up to 10 minutes for each condition: 1) using the Keeogo, 2) using the prescribed knee brace, and 3) using nothing on the knee (optional)
  Walk as far as possible for 6 minutes. Distance in meters and speed in meter/second.
Changes of Timed Up and Go Test results among different conditions | Up to 5 minutes for each condition: 1) using the Keeogo, 2) using the prescribed knee brace, and 3) using nothing on the knee (optional)
  Time in seconds to stand up from a chair, walk 10 feet, turn, walk back to the chair, and sit down.
Changes of 13-Step Stair Test results among different conditions | Up to 10 minutes for each condition: 1) using the Keeogo, 2) using the prescribed knee brace, and 3) using nothing on the knee (optional)
  Ascend and descend a 13-step stair as quickly as possible but safely. Time in seconds till both feet on the top as ascent time. Time in seconds till both feet on the bottom as descent time.
Changes of Pick Up Penny from Floor Test results among different conditions | Up to 3 minutes for each condition: 1) Using the Keeogo; 2) Using the prescribed knee brace; 3) Using nothing on the knee (optional)
  Time in seconds to bend, scoop, lunge, or squat to retrieve a penny from the floor and return to standing. Scored as: not able to perform, perform with physical assistance, perform unassisted
Changes of Short Physical Performance Battery results among different conditions | Up to 15 minutes for each condition: 1) using the Keeogo, 2) using the prescribed knee brace, and 3) Using nothing on the knee (optional)
  Three tests to assess lower extremity functioning: ability to stand for 10 seconds with feet in 3 different positions (together side-by-side, semi-tandem, and tandem), two timed 4-meter walk, and time to rise from a chair five times. Overall score from 0 to 12 with higher score indicating better lower extremity function.

SECONDARY OUTCOMES:
Changes of Numeric Pain Rating Scale results among different conditions | Up to 2 minutes for each condition: 1) using the Keeogo, 2) using the prescribed knee brace, and 3) using nothing on the knee (optional)
  Rate pain on an 11-point numerical scale (0- no pain at all; 10- worst imaginable pain)
System Usability Scale | Up to 5 minutes
  Reliable 10-item scale to evaluate device usability with a 5-point Likert scale from strongly disagree to strongly agree. Overall score from 0 to 100 with higher score indicating better usability.
Usefulness Satisfaction and Ease of Use Questionnaire | Up to 10 minutes
  Reliable 30-item scale to evaluate four dimensions of usability including usefulness, ease of use, ease of learning, and satisfaction with a 7-point Likert scale. Average score from 0 to 7 for each dimension with higher score indicating better usability.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Cardozo, MD, Principal Investigator — James J. Peters Veterans Affairs Medical Center
Locations (1):
- James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mcleod JC, Ward SJ, Hicks AL. Evaluation of the Keeogo Dermoskeleton. Disabil Rehabil Assist Technol. 2019 Jul;14(5):503-512. doi: 10.1080/17483107.2017.1396624. Epub 2017 Nov 2. PMID 29092649
- [Background] McGibbon CA, Sexton A, Jayaraman A, Deems-Dluhy S, Gryfe P, Novak A, Dutta T, Fabara E, Adans-Dester C, Bonato P. Evaluation of the Keeogo exoskeleton for assisting ambulatory activities in people with multiple sclerosis: an open-label, randomized, cross-over trial. J Neuroeng Rehabil. 2018 Dec 12;15(1):117. doi: 10.1186/s12984-018-0468-6. PMID 30541585

DOCUMENTS (1):
  • Informed Consent Form (2024-05-02): https://cdn.clinicaltrials.gov/large-docs/96/NCT04653896/ICF_000.pdf